CLINICAL TRIAL: NCT02885714
Title: ACCURATE Trial - Operative Treatment of Acute Rotator Cuff Tear Related to Trauma; a Placebo-controlled Efficacy Trial
Brief Title: ACCURATE Trial - Operative Treatment of Acute Rotator Cuff Tear Related to Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACCURATE
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Rotator Cuff Tear Related to Trauma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Group I (Placebo Comparator): Placebo surgery + supervised specific exercises
  Interventions: Procedure: Placebo surgery and supervised specific exercises
- Group II (Active Comparator): Rotator cuff repair + supervised specific exercises
  Interventions: Procedure: Rotator cuff repair and supervised specific exercises

INTERVENTIONS:
Procedure: Placebo surgery and supervised specific exercises — The patient is prepared for surgery as normal (plexus+general anesthesia or TIVA, with antibiotic prophylaxis). The arthroscope is introduced in the glenohumeral joint, and thereafter online randomization is performed. The joint space is evaluated. Nothing is to be removed or excised and the use of any vapour or shaver device is not allowed. The presence of a full-thickness rotator cuff tear is verified. Altogether 3 to 5 small stab wounds are made in typical locations resembling locations of typical rotator cuff repair. The time spent in the operating theatre with patients in placebo group should resemble the time spent with patients in the active treatment group and hence give an impression of a rotator cuff repair.
  Arms: Group I
Procedure: Rotator cuff repair and supervised specific exercises — The patient is prepared for surgery as normal (plexus+general anesthesia or TIVA, with antibiotic prophylaxis). The arthroscope is introduced in the glenohumeral joint, and thereafter online randomization is performed. The joint space is evaluated and the presence of a full-thickness rotator cuff tear is verified. The cuff tear is repaired to its anatomic location using suture anchors according to surgeon preference. . A biceps tenotomy or tenodesis may be performed according to surgeon preference if the biceps tendon is noted to be frayed, unstable or inflamed. An additional acromioplasty may be performed according to surgeon preference.
  Arms: Group II

SUMMARY:
Rotator cuff tear is a very common and disabling condition that can be related to acute trauma such as falling on the shoulder. A tear is associated with symptoms such as pain in abduction, abduction weakness and night pain. Rotator cuff tear surgery is a well-established form of treatment in acute rotator cuff tears, although beneficial results have been reported for both conservative and surgical treatment of rotator cuff tears. Rotator cuff tear repair surgery involves a considerable amount of re-ruptures, and it is possible that the repaired tendon do not heal despite surgical repair. On the other hand rotator cuff tears are also found in completely asymptomatic persons and the clinical significance of a rupture may be generally lower than estimated. The above-mentioned factors, as well as recent research and meta-analysis on the treatment of mainly degenerative rotator cuff tears indicate that there is a limited evidence that surgery is not more effective in treating symptomatic rotator cuff tear than conservative treatment alone. However, these previous research findings cannot be applied directly to traumatic tears, although degeneration can be considered always to contribute to the creation of a rotator cuff tear.

During few last decades, despite the lack of evidence on the superiority of one treatment over another, the use of surgery to treat this disorder has been substantially increased. Treatment expectations are found to be important in predicting patient related outcome measures. In addition, surgery itself may produce a profound placebo effect. There are no previous placebo-controlled trials on the topic of interest. In order to find out the true efficacy of surgical treatment of acute, trauma related rotator cuff tears involving mainly the supraspinatus tendon, the investigators have designed this multi-centre, randomized, placebo-controlled efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patient over 45 and below 70 years
2. Acute onset of shoulder symptoms after a traumatic event (any kind of sudden stretch, pull, fall, or impact, on the shoulder that is associated with the onset of symptoms)
3. Shoulder symptoms relating to rotator cuff tear = pain laterally on the shoulder and/or painful motion arc during abduction or flexion
4. MRI documented full thickness supraspinatus (ssp) tear

Exclusion Criteria:

1. Traumatic event of the shoulder due a criminal act of violence with legal consequences
2. A delay of more than 4 months after the onset of symptoms of trauma to the day of intervention
3. Arthroscopically documented partial thickness rotator cuff tear only
4. A large MRI documented full thickness rotator cuff tear, sagittal tear size at the level of footprint larger than 3cm
5. MRI or arthroscopically documented total width of infraspinatus (isp) or subscapularis (ssc) tear
6. MRI or arthroscopically documented fully dislocated biceps tendon (biceps out of the groove) with concomitant subscapularis tear
7. Positive clinical rotatory lag sign (ER1 lag (>10 degrees), lift off lag (involuntary drop against the back), horn blower lag (involuntary internal rotation of the forearm in supported elevated position))
8. Marked fatty degeneration in any of the cuff muscles (more than Fuchs/Goutallier grade 2)
9. Radiographically or MRI documented concomitant fracture line of the involved extremity or bony avulsion of the torn tendon or dislocation of the humeral head or the acromioclavicular joint.
10. Concomitant clinically detectable motoric nerve injury affecting the shoulder
11. Radiographically documented severe osteoarthritis of the glenohumeral joint, Samilson-Prieto 2 or above
12. Non-congruency of the glenohumeral joint in radiographs (Hamada stage 2 or above)
13. Clinical stiffness of the glenohumeral joint (severely limited passive range of motion: glenohumeral external rotation < 30 degrees, and abduction with stabilized scapula <60 degrees)
14. Previous surgery of the affected shoulder (affecting clavicle, scapula or upper third of the humerus)
15. Earlier sonographic or MRI finding of a rotator cuff tear
16. Previous symptoms of the ipsilateral shoulder requiring conservative treatment (glucocorticosteroid injections and/or physiotherapy) delivered by health care professionals during the last five years
17. Systemic glucocorticosteroid or antimetabolite medication during the last 5 years
18. Ongoing treatment for malignancy
19. ASA classification 3 or 4
20. Patient's inability to understand written and spoken Finnish, Norwegian or Swedish
21. History of alcoholism, drug abuse, psychological or other emotional problems likely to jeopardise informed consent
22. Patients with a contraindication/noncomplience for MRI examination or use of electrocautery devices
23. Previous randomization of the contralateral shoulder into the ACCURATE trial
24. Patient's denial for operative treatment and/or participation in the trial

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-12; Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Rotator Cuff index (WORC) compared to baseline at two years. | The change of WORC is also compared to baseline at 3 and 6 months, 1 , 2, 5 and 10 years
  Patient reported disease specific outcome measure for rotator cuff conditions.

SECONDARY OUTCOMES:
Constant Score | 3 and 6 months, 1 , 2, 5 and 10 years
  Shoulder specific outcome measure combining subjective and objective variables
Numeric rating scale of patients' shoulder pain during the last week at rest, during activity and at night. | 3 and 6 months, 1 , 2, 5 and 10 years
  Subjective pain intensity measure. The numeric pain rating scale (pain NRS). Scale 0 to 10. 0 = no pain and 10 = worst possible pain.
15D | 3 and 6 months, 1 , 2, 5 and 10 years
  Generic health-related quality of life instrument
Subjective patient satisfaction | 3 and 6 months, 1 , 2, 5 and 10 years
  Patient reported scale for treatment satisfaction
Rotator cuff integrity in MRI investigation | 2, 5 and 10 years
Development of osteoarthritic signs in radiographs | 2, 5 and 10 years
Development of cuff tear arthropathy in radiographs | 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Juha Kukkonen, MD, PhD, Principal Investigator — Satakunta Central Hospital; Anssi Ryösä, MD, Study Chair — Turku University Hospital; Hanna Björnsson Hallgren, MD, PhD, Study Chair — University Hospital, Linkoeping; Stefan Moosmayer, MD, PhD, Study Chair — Martina Hansens Hospital; Teresa Holmgren, PT, PhD, Study Chair — University Hospital, Linkoeping; Mats Ranebo, MD, Study Chair — Kalmar County Hospital; Berte Bøe, MD, PhD, Study Chair — Oslo University Hospital; Ville Äärimaa, Adj.Prof., Study Director — Turku University Hospital
Locations (17):
- Finland (9):
  - Helsinki University Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Hatanpää Hospital, Tampere
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa
- Norway (4):
  - Sørlandet sykehus HF, Arendal
  - Oslo University Hospital, Ullevål Hospital, Oslo
  - Martina Hansens Hospital, Sandvika
  - St. Olafs Hospital HF, Trondheim
- Sweden (4):
  - Skånevård Sund, Region Skåne, Helsingborg
  - Kalmar County Hospital, Kalmar
  - Linköping University Hospital, Linköping
  - Varberg Hospital, Varberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ryosa A, Kukkonen J, Bjornsson Hallgren HC, Moosmayer S, Holmgren T, Ranebo M, Boe B, Aarimaa V; ACCURATE study group. Acute Cuff Tear Repair Trial (ACCURATE): protocol for a multicentre, randomised, placebo-controlled trial on the efficacy of arthroscopic rotator cuff repair. BMJ Open. 2019 May 19;9(5):e025022. doi: 10.1136/bmjopen-2018-025022. PMID 31110087